CLINICAL TRIAL: NCT05024955
Title: Understanding Shared Decision-Making for Lung Cancer Screening Among Chinese Populations in the U.S.
Brief Title: Evaluating Shared Decision-Making for Lung Cancer Screening Among Chinese Populations in the United States
Status: Withdrawn | Type: Observational
Why Stopped: 0 participants accrued
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0101; NCI-2021-08583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0101 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-18; First posted 2021-08-27 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (interview, discussion): Participants attend an interview over 45-60 minutes and/or a focus group over 1.5 to 2 hours.
  Interventions: Procedure: Discussion; Other: Interview

INTERVENTIONS:
Procedure: Discussion — Attend a focus group
  Other Names: Discuss
Other: Interview — Attend interview

SUMMARY:
This study better understands the views on shared decision-making among Chinese adults who smoke or who have a spouse who smokes. Lung cancer is the second most common cancer among men and women in the United States and is the number one cause of cancer-related mortality among Asians and Pacific Islanders. Clinicians are recommended to initiate conversations about lung cancer screening with eligible patients, provide information about the benefits and harms, and engage in shared decision-making. However, a patient's cultural background can influence decision-making in many ways. Given this, there is a need to understand the perceptions of shared decision-making among different populations (in this case, Asian populations) in order to inform the design of culturally sensitive decision aids for cancer screening. This study evaluates how Chinese populations in the U.S. who currently smoke or who have partners who smoke perceive the process of shared decision-making, their preferences, the perceived barriers and facilitators, and their perspective on currently-available screening tools.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Understand how Chinese populations in the Unites States who currently smoke or who have partners who smoke perceive the process of shared health-related decision-making and their preferences in terms of role involvement, and the barriers to and facilitators of shared decision-making.

II. Evaluate current publicly available lung cancer screening tools from the perspective of Chinese adults who smoke or who have partners who smoke.

OUTLINE:

Participants attend an interview over 45-60 minutes and/or a focus group over 1.5 to 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who self-identify as Chinese
* Live in the U.S. (either citizens or have lived in the U.S. for at least 5 years or more, i.e. long-term residents)
* Age 50-80
* Currently smokes or partner of a person who smokes
* Speak English and/or Mandarin

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are recruited through several sources, including: (1) MD Anderson Cancer Center's (MDACC) Shared Decision Making Core Facility's registry ("REACH" Registry) of patients and caregivers who are willing to participate in decision support development studies (2) community health clinics serving Asian populations in Houston (3) Chinese religious or community groups/centers or at commercial locations catering to the Chinese community (4) social media or virtual groups that cater to Chinese communities of all ages or (5) snowball sampling through referrals from other participants.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
How Chinese populations who smoke or have partners who smoke perceive the process of shared health-related decision-making | through study completion, an average of 1 year
  Data analysis and data collection occurs simultaneously. Data is analyzed using a sequential approach to identify major and minor thematic areas. An initial codebook is developed based on the core questions within the interview guide, the literature, and initial coding of 3-4 transcripts. The internal validity of the codebook is established through detailed discussion between the coders and the research team. The reliability of the codebook is established in the first level of coding (descriptive codes) by double coding 25% of interviews and discussing any discrepancies to reach consensus on codes. Researchers analyze codes to identify the major and minor themes. Findings are summarized and illustrated using verbatim exemplars.
Chinese populations' preferences in terms of role involvement, and the barriers to and facilitators of shared decision-making | through study completion, an average of 1 year
  Data analysis and data collection occurs simultaneously. Data is analyzed using a sequential approach to identify major and minor thematic areas. An initial codebook is developed based on the core questions within the interview guide, the literature, and initial coding of 3-4 transcripts. The internal validity of the codebook is established through detailed discussion between the coders and the research team. The reliability of the codebook is established in the first level of coding (descriptive codes) by double coding 25% of interviews and discussing any discrepancies to reach consensus on codes. Researchers analyze codes to identify the major and minor themes. Findings are summarized and illustrated using verbatim exemplars.
Current publicly available lung cancer screening tools from the perspective of Chinese adults who smoke or who have partners who smoke | through study completion, an average of 1 year
  Data analysis and data collection occur simultaneously. Data is analyzed using thematic analysis. Based on the data from one focus group, an initial codebook is developed based on themes raised by participants. The data is grouped according to broad categories based on the aspects of the tool that the participants provided feedback on, such as: (1) visuals, (2) format of the tool, (3) information, (4) preferences in how risk is presented, (5) decision support, and (6) recommendations for improvement. The codebook is adjusted and refined to include codes that are identified from additional transcripts. Two coders code the transcripts after establishing the codebook's internal validity and reliability through consultation and assistance from other research team members. Findings are summarized and illustrated with verbatim quotes of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Volk, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org